CLINICAL TRIAL: NCT04738344
Title: The Use of Very Long Versus Overlapping Drug Eluting Stents for the Management of Long Coronary Artery Lesions
Brief Title: Very Long Versus Overlapping Stents in Long Coronary Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enough patients enrolled
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIG0122001
Record Dates: First submitted 2020-12-20; First posted 2021-02-04 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease; Chronic Coronary Syndrome; Drug Eluting Stents
Keywords: IVUS; Drug Eluting Stents; Chronic Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous coronary intervention and stent implantation using one long stent (Experimental): Long coronary lesions will be treated percutaneously with a single long stent (more than 40 mm in length) and intravascular ultrasonography (IVUS) will be done immediately after stent deployment to record the baseline picture
  Interventions: Device: Percutaneous Coronary Intervention and Stent Implantation
- Percutaneous coronary intervention and stent implantation using more than one overlapping stents (Experimental): Long coronary lesions will be treated with more than one overlapping stents and intravascular ultrasonography (IVUS) will be done immediately after stent deployment to record the baseline picture
  Interventions: Device: Percutaneous Coronary Intervention and Stent Implantation

INTERVENTIONS:
Device: Percutaneous Coronary Intervention and Stent Implantation — Percutaneous Coronary Intervention and Stent Implantation will be implanted as recommended by guidelines and according to the standard techniques.
  Other Names: PCI

SUMMARY:
This study is performed to compare the angiographic and clinical outcomes of the use of single long stent versus overlapping stents in the treatment of long coronary lesions in patients with chronic coronary syndrome.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) in diffuse coronary artery disease is still considered a big obstacle for interventional cardiologists. Very long coronary lesions are usually found, and implantation of a single stent was a great problem forcing the operator to do overlapping of several stents.

Recently, new stent designs with increasing length are developed and emerging as a great tool for the percutaneous treatment of long lesions. Nowadays, stents up to 60 mm are available to be used in these cases reducing stent overlap.

Intravascular ultrasound (IVUS)-guided percutaneous coronary intervention has been shown in clinical trials, registries, and meta-analyses to be associated with a reduction in clinical events after percutaneous coronary intervention; however, IVUS utilization during percutaneous coronary intervention remains low in the United States and worldwide. The impact of IVUS in these complex lesions may be associated with a lower rate of clinical adverse events in comparison with angiography alone.

The study will be conducted on forty patients with chronic stable angina on maximal medical treatment who are going to have elective coronary angiography and elective PCI and having one long coronary lesion that is more than 40 mm in length, they will be randomized into either treatment of the lesion with a single very long stent (more than 40 mm in length) or with more than one overlapping stents in 1:1 randomization. Control angiography and IVUS will be done to the 2 groups after 6 months and the major cardiovascular outcomes will be addressed at 1,3 and 6 months follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Single vessel disease and undergoing PCI for significant long lesion.
* Chronic stable angina on maximal medical treatment.

Exclusion Criteria:

* Patients presenting with acute coronary syndromes.
* Patients having two or more vessel disease on coronary angiography.
* Previous myocardial infarction.
* Previous vascularization either by PCI or bypass grafting.
* Very low ejection fraction less than 35%.
* Renally impaired patients with Creatinine clearance less than 50 ml/min.
* Contraindication to dual antiplatelet drug therapy.
* Contraindication to coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Coronary angiographic criteria after 6 months of stent deployment | 6 months
  Number of participants with any form in-stent restenosis using control coronary angiography at 6 months
(IVUS) after 6 months of stent deployment | 6 months
  Number of participants with any form in-stent restenosis using Intravascular Ultrasonography (IVUS) at 6 months to assess subclinical neointimal proliferation and in-stent restenosis
Major Cardiovascular and Cerebrovascular Events (MACCE) after 6 months | 6 months
  Number of patients with any Major Cardiovascular and Cerebrovascular Events (MACCE) at 6 months of stent deployment

SECONDARY OUTCOMES:
Any Major Bleeding Event | 6 months
  Number of patients with Any Major Bleeding Event as defined by the International Society of Thrombosis and Haemostasis (fatal bleeding, and/or symptomatic bleeding in a critical organ or area, and/or bleeding causing a fall in hemoglobin level of ≥ 2 g/dl or 1.24 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Sobhy, MD, Study Chair — University of Alexandria - Egypt; Amr Zaky, MD, Study Director — University of Alexandria - Egypt; Ahmed M El Amrawy, MD, Principal Investigator — University of Alexandria - Egypt
Locations (2):
- Egypt (2):
  - University of Alexandria, Alexandria
  - International Cardiac Center (ICC), Alexandria

IPD SHARING:
Plan to Share IPD: No
IPD may be shared with researchers if requested